CLINICAL TRIAL: NCT00312052
Title: A Randomized, Double-Blind, Placebo-Controlled Study of the Safety and Tolerability of E5555, and Its Effects on Markers of Intravascular Inflammation in Subjects With Coronary Artery Disease
Brief Title: Safety and Tolerability of E5555 and Its Effects on Markers of Intravascular Inflammation in Subjects With Coronary Artery Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: E5555-G000-201; 2005-006029-94 (EudraCT Number)
Record Dates: First submitted 2006-04-05; First posted 2006-04-07 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-11

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — E 5555

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- E5555 50 mg (Experimental): Participants received one 50 mg E5555 and two 100 mg placebo tablets, once orally daily for 24 weeks.
  Interventions: Drug: E5555; Drug: Placebo
- E5555 100 mg (Experimental): Participants received one 50 mg placebo, one 100 mg E5555 and one 100 mg placebo tablets, once orally daily for 24 weeks.
  Interventions: Drug: E5555; Drug: Placebo
- E5555 200 mg (Active Comparator): Participants received one 50 mg placebo and two 100 mg E5555 tablets were taken orally once daily for 24 weeks.
  Interventions: Drug: E5555; Drug: Placebo
- Placebo (Placebo Comparator): Participants received one 50 mg placebo and two 100 mg placebo tablets, once orally daily for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: E5555 — 50 mg or 100 mg E5555 tablets
  Arms: E5555 100 mg; E5555 200 mg; E5555 50 mg
Drug: Placebo — 50 mg and/or 100 mg placebo tablets

SUMMARY:
The primary purpose of this study is to assess the safety and tolerability of E5555 in subjects with coronary artery disease.

DETAILED DESCRIPTION:
This was a multicenter, randomized, double-blind, placebo-controlled trial of E5555, a PAR-1 inhibitor. The total duration of individual study participation was 28 weeks (196 days). This included a treatment period of 24 weeks (168 days) and a follow-up period of 4 weeks (28 days).

ELIGIBILITY:
INCLUSION CRITERIA:

1. Males or Females, 45 - 80 years of age
2. Confirmed coronary artery disease defined as one of the following:

   * Post-acute coronary syndrome or myocardial infarction or
   * Post percutaneous coronary intervention or coronary artery bypass graft or oAngina pectoris with documented (electrocardiogram or imaging study) ischemia or
   * Angiographically documented lesion occluding ≥70% of a coronary vessel

   And at high risk as defined as one or more of the following:
   * Elevated hsCRP (high-sensitivity C-reactive protein)
   * Diabetes mellitus
   * History of carotid artery disease and/or peripheral artery disease
   * Thrombo-embolic transient ischemic attack or stroke >1 year prior to screening
3. All subjects must be receiving low dose aspirin and/or clopidogrel and/or ticlopidine.

EXCLUSION CRITERIA

1. History of acquired or congenital bleeding disorder, coagulopathy or platelet disorder, or history of pathological bleeding within the last 6 months
2. History of intracranial bleeding, history of hemorrhagic retinopathy or known structural cerebral vascular lesion
3. Clinically significant hematological, hepatic or renal abnormalities
4. Patients with some specific ST-segment changes, severe congestive heart failure or uncontrolled cardiac arrhythmias at baseline
5. Recent significant (as determined by the investigator) cardiovascular events

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Actual)
Dates: Start 2007-09; Primary Completion 2008-03 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability - especially the risk of bleeding | 6 months

SECONDARY OUTCOMES:
Incidence of major adverse cardiovascular events; the effect on platelet aggregation inhibition. Exploratory Outcome Measure: effects on endovascular inflammatory processes | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: John Riefler, MD, Study Director — Eisai Limited
Locations (2):
- United States (2):
  - Florida Research Network, Gainesville, Florida
  - Great Lakes Heart Center of Alpena, Alpena, Michigan

REFERENCES:
- [Derived] Wiviott SD, Flather MD, O'Donoghue ML, Goto S, Fitzgerald DJ, Cura F, Aylward P, Guetta V, Dudek D, Contant CF, Angiolillo DJ, Bhatt DL; LANCELOT-CAD Investigators. Randomized trial of atopaxar in the treatment of patients with coronary artery disease: the lessons from antagonizing the cellular effect of Thrombin-Coronary Artery Disease Trial. Circulation. 2011 May 3;123(17):1854-63. doi: 10.1161/CIRCULATIONAHA.110.001404. Epub 2011 Apr 18. PMID 21502571